CLINICAL TRIAL: NCT05994248
Title: Absorbable and Synthetic Mesh: A Multicenter, Prospective, Non-Inferior, Randomized Controlled Trial
Brief Title: Randomized Controlled Trial (RCT) Umbilical Hernia Repair (UHR) Absorbable vs Non-absorbable Synthetic Mesh
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study was never opened and PI now leaving institution
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00097688
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-05

CONDITIONS: Umbilical Hernia
Keywords: Randomized Controlled Trial (RCT); Absorbable Mesh; Non-Absorbable Mesh
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Non-Absorbable Synthetic Mesh (Experimental): Subjects randomized to the non-absorbable synthetic mesh arm will undergo the procedure (umbilical hernia repair) to receive Marlex mesh.
  Interventions: Device: Marlex
- Absorbable Synthetic Mesh (Active Comparator): Subjects randomized to the absorbable synthetic mesh arm will undergo the procedure (umbilical hernia repair) to receive Enform mesh.
  Interventions: Device: Enform Mesh

INTERVENTIONS:
Device: Enform Mesh — Use of absorbable mesh in umbilical hernia repair
  Arms: Absorbable Synthetic Mesh
Device: Marlex — Use of non-absorbable mesh in umbilical hernia repair
  Arms: Non-Absorbable Synthetic Mesh

SUMMARY:
The goal of this study is to see which of two types of mesh is better for fixing an umbilical hernia. One type of mesh is an absorbable synthetic mesh, which goes away on its own in the body, and the other type of mesh is a non-absorbable mesh, which stays in the body forever. The researchers will check if the hernia comes back, how it affects the patient's quality of life, and if there are any problems after the surgery during a three-year period.

DETAILED DESCRIPTION:
The goal of this study is to compare the use of absorbable synthetic (AS) mesh versus non-absorbable mesh (NAS) mesh to determine the 3-year recurrence, quality of life (QOL) and postoperative complications in umbilical hernia repair. Patients will be randomized into one of two arms to receive an absorbable (Enform) mesh or non-absorbable (Marlex) mesh. Patients will undergo an umbilical hernia repair with the mesh assigned to their randomization cohort. The hernia recurrence, quality of life and postoperative outcomes to determine if the two meshes are non-inferior.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Primary umbilical hernia repair (UHR) [as defined by European Hernia Society (EHS) guidelines primary midline abdominal wall defect from 3 cm above to 3 cm below the umbilicus]
* Undergoing elective laparoscopic or open repair
* Defect size of 1-4cm2
* Centers for Disease Control and Prevention (CDC) class 1 & 2 wounds

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Umbilical Hernia Recurrence | 3-years postoperatively
  The rate of hernia recurrence 3-years postoperatively

SECONDARY OUTCOMES:
Mesh Related Complication - Mesh infection | 1-year postoperatively
  The rate of mesh infection within 1-year postoperatively
Mesh Related Complication - Mesh excision | 1-year postoperatively
  The rate of mesh excision within 1-year postoperatively
Postoperative Outcome - 30-day readmission | 30-days postoperatively
  The rate of 30-day readmission
Postoperative Outcome - Seroma | 3-years postoperatively
  The rate seroma within 3-years postoperatively
Postoperative Outcome - Hematoma | 3-years postoperatively
  The rate of hematoma within 3-years postoperatively
Postoperative Outcomes - Intra-abdominal abscess | 3-years postoperatively
  The rate of intra-abdominal abscess within 3-years postoperatively
Postoperative Outcome - Wound cellulitis | 3-years postoperatively
  The rate of wound cellulitis within 3-years postoperatively
Postoperative Outcome - Wound infection | 3-years postoperatively
  The rate of wound infection within 3-years postoperatively
Postoperative Outcome - Superficial wound breakdown | 3-years postoperatively
  The rate of superficial wound breakdown within 3-years postoperatively
Postoperative Outcomes - Mortality | 3-years postoperatively
  The rate of mortality within 3-years postoperatively
Postoperative Outcomes - Length of stay | 3-years postoperatively
  The length of stay (LOS) in the hospital postoperatively
Quality of Life (QOL) | 3-years postoperatively
  QOL within 3-years of surgery as measured by the Carolinas Comfort Scale (CCS), a validated hernia specific QOL questionnaire. The CCS has 23 questions across 3 domains (mesh sensation, pain, and movement) that are scored 0-5 and N/A. Higher scores indicate worse symptoms. A score of 2 or more in any category is considered "symptomatic"; a score of 0 or 1 is considered "asymptomatic". Data will be reported as the frequency and percentage of "symptomatic" or "asymptomatic" for each of the 3 domains.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Heniford, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to other researchers.